CLINICAL TRIAL: NCT07097038
Title: Analgesic Effect and Safety of Oliceridine and Oxycodone in Vitrectomy: a Randomized Controlled Trial
Brief Title: Analgesic Effect and Safety of Oliceridine and Oxycodone in Vitrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HenanPPH-FNN2
Record Dates: First submitted 2025-07-22; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Vitrectomy
Keywords: Basic anesthesia
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine group (Experimental): Intraoperative analgesia: Oliceridine 0.015mg/kg
  Interventions: Drug: Oliceridine
- Oxycodone group (Active Comparator): Intraoperative analgesia oxycodone 0.04mg/kg
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oliceridine — Intraoperative analgesia should be administered with Oliceridine
  Arms: Oliceridine group
Drug: Oxycodone — Oxycodone is used for intraoperative analgesia
  Arms: Oxycodone group

SUMMARY:
Traditional opioid analgesia is a method to treat moderate to severe pain. However, the use of opioids is not without risks. When treating acute pain, patients may have hypotension, respiratory depression, hypoxia, nausea and vomiting, irritability and pruritus. The aim of this study was to evaluate the analgesic effect and safety of g-protein-biased μ - opioid receptor agonists Oliceridine and oxycodone in vitrectomy.

DETAILED DESCRIPTION:
a total of 120 patients scheduled for vitrectomy were randomly divided into Oliceridine group (n = 60) and oxycodone group (n = 60). The main outcome measure was visual analogue scale (VAS) at 2 hours after operation, and the secondary outcome measures included intraoperative analgesic drug addition, VAS scores at 6 and 24 hours after operation, respiratory depression (oxygen saturation < 90%) and incidence of adverse reactions (nausea, vomiting, dizziness).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, ASA Ⅰ - Ⅱ (the age of patients with vitreous surgery can be relaxed to 75 years old, and serious systemic diseases need to be excluded);
* Vitrectomy with local anesthesia (retrobulbar / peribulbar block) combined with intravenous sedation and analgesia (such as maculopathy, retinal detachment, etc.);
* Preoperative VAS score ≤ 3, can cooperate with pain and sedation score;
* Signed informed consent.

Exclusion Criteria:

* Be allergic to test drugs or opioids, or have a history of opioid abuse;
* Severe cardiopulmonary disease (such as heart failure, COPD), liver and kidney dysfunction (alt/ast > 3 times normal, creatinine > 177 μ mol/l);
* Glaucoma (avoiding the risk of fluctuation of intraocular pressure), sinus bradycardia (< 50 beats / min, preventing aggravation of oculo cardiac reflex);
* Used analgesic / sedative drugs within 24 hours before surgery;
* Those who are unable to cooperate due to mental illness or cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
VAS score 2 hours after operation | From enrollment to the end of treatment at 1 day
  Postoperative 2-hour VAS score (total score of 10, 0 indicates no pain, and 10 indicates the most severe unbearable pain)

SECONDARY OUTCOMES:
Adverse reactions | From enrollment to the end of treatment at 1 day
  ncidence of nausea, vomiting, dizziness, headache, constipation, itching, and hypoxia

IPD SHARING:
Plan to Share IPD: No